CLINICAL TRIAL: NCT06460532
Title: Effects of Diaphragm Manual Therapy Versus Sustained Natural Apophyseal Glide on Pain, Range of Motion and Functional Disability in Patients With Mechanical Neck Pain
Brief Title: Effects of Diaphragm Manual Therapy Verses Sustained Natural Apophyseal Glide in Mechanical Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0196 Anam
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Neck Pain
Keywords: disability; muscle strength; pain; Range of Motion
MeSH Terms: conditions — Neck Pain; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Diaphragm Manual Therapy (Experimental): Group A were receiving diaphragm Manual therapy by Leon Chaitow. Subsequently, in order to indirectly stretch and mobilize the fibres of the diaphragm, diaphragmatic manual therapy was used, which should result in improved muscle contraction and reduced tension. The doming diaphragmatic technique and the manual diaphragmatic release technique, both as described by Leon Chaitow, will be among the experimental methods employed. For 10 min, both manoeuvres were performed in 2 sets of 10 repetitions each, separated by 1 min.
  Interventions: Other: Baseline treatment
- Group B: Sustained Natural Apophyseal Glide (SNAGs) (Active Comparator): Group B has received the Sustained natural apophyseal glide (SNAGS). Treatment procedure for SNAGs was sustained natural apophyseal glides whereby the patient attempts to actively move a painful or stiff joint through its ROM while the therapist overlays an accessory glide parallel with the treatment plane. SNAG mobilization was given to a patient (as defined by Mulligan) sitting on a chair. At the same time, the treating physiotherapist stood behind by placing the medial border of the distal phalanx of the thumb on the spine of one vertebra above the affected region. The glides were given with the tip of the thumb placed at an angle of 45° along the eyeball direction reinforced by another thumb. In the session, glides were repeated six times, and three sets were given at C3-C7 cervical levels.
  Interventions: Other: Baseline treatment

INTERVENTIONS:
Other: Baseline treatment — Transcutaneous Electric Nerve Stimulation (TENS) of Care Vision company will be applied, with a pulse duration of 250 microseconds at a frequency of 80 Hz for 15 min in the suboccipital region and the trapezius bilaterally.

SUMMARY:
Mechanical neck pain is defined as pain and discomfort localized between the superior nuchal line, cervical spine, and the spinous process of the first thoracic vertebra. Some of the most typical factors include continuous use of mobile phones and computers, working in sedentary jobs, etc. Study aimed to compare diaphragm manual therapy and Sustained Natural Apophyseal Glide on pain, range of motion and functional disability in patients with mechanical neck pain.

DETAILED DESCRIPTION:
This project will be a Randomized Clinical Trial conducted to check the effects of Diaphragm manual therapy versus sustained natural apophyseal glide on pain, range of motion and functional disability in patients with mechanical neck pain at Sehat Medical Complex Lahore through non-probability convenient sampling technique on 34 patients will be allocated using simple random sampling through Computer generated Randomization into Group A and Group B. Group A will be treated with Diaphragm Manual Therapy and baseline treatment was given and Group B with Sustained Natural Apophyseal Glide and baseline treatment was given. All Exercise were performed 3 times a week for total 4 weeks. Outcome measures will be conducted through NPRS for pain, ROM measured by Goniometer, and Neck Disability Index (NDI) for Disability after 4 weeks. Data was analyzed during SPSS software version 25. After assessing the normality of data by the Shapiro-Wilk test, it decided whether either parametric or non-parametric tests were used within a group or between two groups.

ELIGIBILITY:
Inclusion Criteria:

* Age group between 18 and 40 years
* Both gender male and female
* Individuals having localized pain or stiffness in the cervical spine or both combined between C3 and C7 without upper-limb radiculopathy
* Pain reported on NPRS score ˃3 to <7/10 in neck region for more than 3 months.
* Limited Neck ROM
* Negative Spurling's test, traction test, upper limb tension test, and shoulder abduction test

Exclusion Criteria:

Patients were excluded if they were diagnosed with the following conditions for ˃6 months

* Tuberculosis, carcinoma, heart disease, and osteoporosis
* Neural disorders due to prolapsed intervertebral disc
* Any trauma or localized infection in neck region
* Upper motor neuron disease, cervical stenosis, and metabolic diseases in bone and joint
* Hyper flexibility
* Open sores
* Ongoing radiotherapy, chemotherapy, steroid therapy, or anticoagulants
* Psychiatric diseases such as phobia/obsession and depression
* Allergy to hot pack
* Patients with history of surgery in cervical spine region with in a year.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2024-06-30 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | upto 4 weeks
  The primary outcome was pain assessment by the Numeric Pain Rating Scale (NPRS). This is a reliable self-reported 11-point numeric scale, where each number reflects the intensity of the pain referred by the patient: "0" stands for "no pain" and "10" for "the worst possible pain". Patients verbally selected 3 values that were most in line with the intensity of pain that they had experienced in the previous 24 h, corresponding to current pain and to his/her best and worst pain. The average of the 3 ratings was used to represent the patient's level of pain over the previous 24 h. NPRS was assessed before and after each treatment session. The reliability is (r = 0.96 and 0.95, respectively) and validity correlations range from 0.86 to 0.95
Neck disability Index (NDI) | upto 4 weeks
  Disability was assessed using the Urdu version of the Neck Disability Index (NDI). This is a reliable scale and was self-assessed by the patients and filled in at the beginning and at the end of the whole treatment. The results of this questionnaire have been utilized to evaluate the disability. It consists of 10 items: 7 linked to activities of daily living, 2 to pain, and 1 to concentration. From 0 to 5, each item received a score. Higher scores corresponded to more disability, and the total score was reported as a percentage. The reliability is between 0.50 and 0.98.
Universal Goniometer | upto 4 weeks
  An instrument called a goniometer was used to measure a joint's range of motion. Physical therapists typically use a goniometer to measure a range of motion. At the initial evaluation, the therapist can determine the possible range of motion using a goniometer. The reliability is (r = .58). Neck ROM will be measured in this study using a Universal Goniometer.

CONTACTS AND LOCATIONS:
Overall Officials: Anam Akram, MSPT*, Principal Investigator — Riphah International University,Lahore; samrood Akram, Study Director — Riphah International University
Locations (1):
- Sehat Medical Complex, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saleem I, Zahoor IA, Rana AA, Sarfraz S, Ibrahim M, Ghaffar N. Comparison of Sustained Natural Apophyseal Glide and Natural Apophyseal Glide Effects on Pain, Range of Motion and Neck Disability in Patients with Chronic Neck Pain: Comparison of Sustained Natural Apophyseal Glide and Natural Apophyseal Glide Effects. Pakistan Journal of Health Sciences. 2022:154-8.
- [Background] Tatsios PI, Grammatopoulou E, Dimitriadis Z, Koumantakis GA. The Effectiveness of Manual Therapy in the Cervical Spine and Diaphragm, in Combination with Breathing Reeducation Exercises, in Patients with Non-Specific Chronic Neck Pain: Protocol for Development of Outcome Measures and a Randomized Controlled Trial. Diagnostics (Basel). 2022 Nov 4;12(11):2690. doi: 10.3390/diagnostics12112690. PMID 36359533
- [Background] Pal A, Misra A. EFFECTIVENESS OF SNAG MOBILIZATION ON COMPUTER PROFES-SIONALS WITH MECHANICAL NECK PAIN AND MOBILITY DEFICIT. Int J Physiother Res. 2019;7(2):3022-27.
- [Background] Haghighat F, Moradi R, Rezaie M, Yarahmadi N, Ghaffarnejad F. Added Value of Diaphragm Myofascial Release on Forward Head Posture and Chest Expansion in Patients With Neck Pain: A Randomized Controlled Trial. 2020.
- [Background] Simoni G, Bozzolan M, Bonnini S, Grassi A, Zucchini A, Mazzanti C, Oliva D, Caterino F, Gallo A, Da Roit M. Effectiveness of standard cervical physiotherapy plus diaphragm manual therapy on pain in patients with chronic neck pain: A randomized controlled trial. J Bodyw Mov Ther. 2021 Apr;26:481-491. doi: 10.1016/j.jbmt.2020.12.032. Epub 2021 Feb 16. PMID 33992285
- [Background] Jabbar KM, Gandomi F. The comparison of two corrective exercise approaches for hyperkyphosis and forward head posture: A quasi-experimental study. J Back Musculoskelet Rehabil. 2021;34(4):677-687. doi: 10.3233/BMR-200160. PMID 33896809
- [Background] Bernal-Utrera C, Gonzalez-Gerez JJ, Anarte-Lazo E, Rodriguez-Blanco C. Manual therapy versus therapeutic exercise in non-specific chronic neck pain: a randomized controlled trial. Trials. 2020 Jul 28;21(1):682. doi: 10.1186/s13063-020-04610-w. PMID 32723399